CLINICAL TRIAL: NCT00494429
Title: Optimizing Pain Treatment in Pre-Term Neonates
Brief Title: Optimizing the Use of Morphine in Pre-Term Neonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John van den Anker (Other)
Collaborators: University of Louisville (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor-Investigator, John van den Anker, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPRU-10750; Inulin IND #73093
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Premature Neonates
Keywords: Preterm Neonates; Morphine; Critically ill
MeSH Terms: conditions — Critical Illness | interventions — Morphine; Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Gestational Age< 29 weeks will be administered a loading dose of 0.05 mg/kg I.V. morphine over 30-minutes, followed by a continuous infusion of 0.005 mg/kg/hr.
  Interventions: Drug: Morphine
- 2 (Experimental): Gestational Age>= 29 weeks will be administered a loading dose of 0.1 mg/kg I.V. morphine over 30-minutes, followed by a continuous infusion of 0.01 mg/kg/h.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Gestational Age< 29 weeks: A loading dose of 0.05 mg/kg I.V. morphine over 30-minutes, followed by a continuous infusion of 0.005 mg/kg/h.
  Other Names: inulin
  Arms: 1
Drug: Morphine — Gestational Age>= 29 weeks: A loading dose of 0.1 mg/kg I.V. morphine over 30-minutes, followed by a continuous infusion of 0.01 mg/kg/h.
  Other Names: Inulin
  Arms: 2

SUMMARY:
The purpose of this study is to improve the dosing of morphine in critically ill premature neonates.

DETAILED DESCRIPTION:
The investigators hypothesize that identifying co-variates predictive of variability in morphine disposition and/or response will provide the scientific basis for rationale and individualized morphine dosing schemes in neonates and young infants.

60 preterm neonates ranging in gestational age from 22 to 32 weeks will be recruited from the NICU. Stratification by gestational age will be done to ensure broad representation. The decision to initiate morphine therapy will be based solely on clinical indications. Prior to morphine dosing, a biochemical assessment of hepatic and renal function will be obtained. A 0.05 mg/kg loading dose of morphine will be given by an intravenous infusion over 30-minutes in preterm neonates with a gestational age of less than 29 weeks, followed by a continuous infusion of 0.005 mg/kg/h, whereas a loading dose of 0.1 mg/kg will be given in preterm neonates with a gestational age of 29 weeks or more followed by a continuous infusion of 0.01 mg/kg/h. Pain assessment will be performed at baseline (prior to study medication administration) and at .5, 1, 2, 4, 8, 12 and 24 hours after the dose. At each of these time points infants will be videotaped for two minutes with two cameras. Videotapes will be scored afterward using standard validated pain assessment tools for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates of both genders and all races
* postnatal age less than 30 days
* an indwelling (peripheral or umbilical) arterial line, and
* a clinical indication for intravenous morphine administration

Exclusion Criteria:

* Neonates with severe asphyxia, grade III or IV intraventricular hemorrhage, major congenital malformations/facial malformations, neurological disorders, and those receiving continuous or intermittent neuromuscular blockers.
* clinical or biochemical evidence of hepatic and renal compromise (including systemic hypoperfusion) or
* received drugs that are UGT2B7 substrates (including Lorazepam, ibuprofen, valproic acid, naloxone and other morphine derivatives or propanolol)

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2005-05; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety: Infants will have continuous monitoring of vital signs, oxygen saturation, movements and adverse events to determine the safety of morphine. | study duration
Pharmacodynamics: The Neonatal Infant Pain (NIP) and Premature Infant Pain Profile (PIPP) will be performed at baseline, (prior to drug administration)and at pre-determined time intervals after the dose to assess pain for the efficacy of morphine. | study duration
Pharmacokinetics: The concentrations of morphine and its metabolites will be measured in plasma and urine at pre-determined time points and will be used to calculate the formation and elimination clearances of morphine and its metabolites. | study duration
Pharmacogenetics: Impact of genetic variation in the UGT2B7 gene on the formation clearances of the morphine metabolites will be studied as well as the genetic variation in the µ-opioid receptor, COMT, and β-arrestin 2 genes on the PD of morphine use | study duration

CONTACTS AND LOCATIONS:
Overall Officials: John N. van den Anker, M.D., Ph.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States